CLINICAL TRIAL: NCT01399060
Title: Cough and Taste Preferences in Adolescents and Adults
Brief Title: Cough Sensitivity and Taste Preferences
Acronym: CAP
Status: Completed | Type: Observational
Sponsor: Monell Chemical Senses Center (Other)
Collaborators: Pennsylvania Department of Health (Other Government)
Responsible Party: Principal Investigator, Julie A. Mennella, Member, Monell Chemical Senses Center
Other Study IDs: 812923; SAP No. 4100054860 (Other Grant/Funding Number: Pennsylvania Department of Health)
Record Dates: First submitted 2011-07-19; First posted 2011-07-21 (Estimated); Last update posted 2013-10-24 (Estimated); Status verified 2013-10

CONDITIONS: Smoking
Keywords: Cough; tobacco smoke exposure
MeSH Terms: conditions — Smoking; Cough

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Saliva samples will be obtained from the subjects, if consented. These saliva samples will be genotyped at the Monell Center for genes that may play a role in chemical irritation and flavor-perception. This testing is exploratory in nature.
Oversight: Data Monitoring Committee: No

SUMMARY:
This single-site, within-subject, experimental study is designed to test the hypothesis children who live in a household in which one or both of their parent smoke will exhibit a higher cough threshold and will prefer more intense sweet tastes than children who live in a household where neither parent smokes. Subjects will include at least 50 racially and ethnically diverse, healthy children aged 10 to 17 years (a critical time for experimenting with tobacco) and a parent. The sample will comprise two groups: Non-Environmental Tobacco Smoke (ETS) Exposed (neither the child nor parents has ever smoked or been exposed to environmental tobacco smoke (ETS) in the home), and ETS-Exposed (the parent has smoked at least 3 cigarettes per day for at least five years in the home, with the child living in the home continuously). Cough sensitivity will be measured using a standard single-inhalation challenge, a test of the minimum concentration of capsaicin (the spicy chemical in hot peppers) needed to elicit cough. Sweet taste preferences will be measured using a forced-choice paired comparison method of liquids which differ in sucrose content. Measures of breath carbon monoxide will validate the smoking status of parents and their adolescent children. The key comparison will be between Non-ETS Exposed and ETS-Exposed children, with the difference between smoking and non-smoking parents as a positive control. Because smoking and non-smoking families may differ in ways besides tobacco exposure, the investigators will obtain health histories (with a focus on respiratory illness), smoking histories, measures of body weight, diet, and responses to personality tests (including susceptibility to addiction). The investigators will also obtain genomic DNA from saliva samples. Genes for chemosensory receptors that are part of the cough reflex pathway and genotype may account for aspects of cough sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults and children of both genders will be studied.
* Ages of children will range from 10 to 17 years.

Exclusion Criteria:

* Subjects with a current respiratory illness of any type (including current infection or infection within the last month, asthma, chronic obstructive pulmonary disease, bronchitis of any type, or any other breathing issue).
* Subjects who report that they have a history of asthma or other chronic respiratory condition.
* Subjects who report unusual sensitivity to environmental odors (e.g., reactive airways, multiple chemical sensitivity).
* Subjects who report that they have a history or allergic reactions to foods and/or chemicals.
* Subject who report that they are diabetic, or on any medication, with exception of birth control pills (for mothers only).

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Approximately 50 parent-child dyads (N=100 subjects total) will be tested on two days separated by at least 2-3 days. The children will be between the ages of 10 and 17 years. Half of sample will be children whose mothers are current smokers and the other have will be children whose mothers and fathers never smoked in their lifetimes.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2011-04; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
cough threshold | 90 minutes
  Cough threshold (sensitivity) will be measured using a standard single-inhalation challenge, a test of the minimum concentration of capsaicin (the spicy chemical in hot peppers) needed to elicit cough

SECONDARY OUTCOMES:
smoking history (of parents) | 10 minutes
  We will determine the smoking history of the parent via questionnaires to examine the relationship between cough threshold and smoking history of parent for both children and parent
Genotype | One year
  We will genotype saliva samples for genes for chemosensory receptors that are part of the cough reflex pathway and genotype to explore individual differences in cough sensitivity

CONTACTS AND LOCATIONS:
Overall Officials: Julie A. Mennella, PhD, Principal Investigator — Monell Chemical Senses Center; Paul Wise, PhD, Principal Investigator — Monell Chemical Senses Center
Locations (1):
- Monell Chemical Senses Center, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Result] Wise PM, Mennella JA, Finkbeiner S. Impaired cough sensitivity in children of smokers. Nicotine Tob Res. 2013 Feb;15(2):603-7. doi: 10.1093/ntr/nts198. Epub 2012 Aug 17. PMID 22904107